CLINICAL TRIAL: NCT00598078
Title: Multiple-dose, Double-blind, Placebo-controlled, Crossover Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Sodium Oxybate (Xyrem) in Subjects With Moderate to Severe Essential Tremor
Brief Title: Multiple-dose,Double-blind,Placebo-controlled Study of Sodium Oxybate in Patients With Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06-015
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2011-12

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Sodium Oxybate
- 2 (Experimental)
  Interventions: Drug: Sodium Oxybate
- 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium Oxybate — Dose 1
  Arms: 1
Drug: Sodium Oxybate — Dose 2
  Arms: 2
Other: Placebo — Dose 3
  Arms: 3

SUMMARY:
To determine the relationship between drug plasma levels and safety, tolerability and efficacy in patients with essential tremors after dosing with Sodium oxybate

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate or severe classic essential tremor (bilateral, largely symmetric postural or kinetic tremor involving hands and forearms.
* Willingness to abstain from ethanol and caffeine intake for at least 48 hours prior to Days 1 and 4 and on inpatient days

Exclusion Criteria:

* Subjects with a clinically significant unstable medical abnormality, chronic disease or history or presence of significant hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, psychiatric, or metabolic disease or any other abnormality
* Subjects who are on sodium-restricted diets
* Subjects with a known history of sleep apnea

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Ellenbogen, DO, Principal Investigator — Quest Research Institute
Locations (1):
- Quest Research Institiute, Bingham Farms, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A, Then B, Then C: Day 1: Sodium Oxybate 0.75g at ~8am, Sodium Oxybate 0.75g at ~10am, placebo at ~12pm; Day 2:Sodium Oxybate 1.5g at ~8am, placebo at ~10am, Sodium Oxybate 1.5g at ~12pm; Day 3:Placebo at ~8am, ~10am, and ~12pm
- Regimen A, Then C, Then B: Day 1: Sodium Oxybate 0.75g at ~8am, Sodium Oxybate 0.75g at ~10am, placebo at ~12pm; Day 2: Placebo at ~8am, ~10am, and ~12pm; Day 3: Sodium Oxybate 1.5g at ~8am, placebo at ~10am, Sodium Oxybate 1.5g at ~12pm;
Period: Period 1 (Day 1)
Arm/Group | Regimen A, Then B, Then C | Regimen A, Then C, Then B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2 (Day 2)
Arm/Group | Regimen A, Then B, Then C | Regimen A, Then C, Then B
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 3 (Day 3)
Arm/Group | Regimen A, Then B, Then C | Regimen A, Then C, Then B
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All treated study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 60.0 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Modified FTM(Fahn-Tolosa-Marin) Essentials Tremor Rating Scale, Sum of All Essential Rating Tremor Scales Including Voice Tremor
Description: The modified FTM sum of all essential rating tremor scales including voice tremor includes: the tremor rating taken for the left & right hands individually at rest, with posture (arms outstretched), with action (finger to nose). It also includes an evaluation of voice with scores for AAA & EEE sounds, an action evaluation of left & right hands pouring, bringing liquids to mouth, drawing large & small spirals. Scores for indiviuals items range from 0 (no tremor) to 4 (severe tremor). The sum ranges from 0 (no tremor) to 72 points (higher amplitude/more tremors).
Time Frame: Hour 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Points
Groups:
- Sodium Oxybate 1.5 Grams (A): Sodium Oxybate 0.75g at ~8am, Sodium Oxybate 0.75g at ~10am, placebo at ~12pm (Day 1 only)
- Sodium Oxybate 3 Grams (B): Sodium Oxybate 1.5g at ~8am, placebo at ~10am, Sodium Oxybate 1.5g at ~12pm (Day 2 or 3)
- Placebo (C): Placebo at ~8am, ~10am, and ~12pm (Day 2 or 3)
Arm/Group | Sodium Oxybate 1.5 Grams (A) | Sodium Oxybate 3 Grams (B) | Placebo (C)
Number analyzed (Participants) | 20 | 20 | 19
Points | 13.4 [9.05 to 17.65] | 10.8 [6.50 to 15.10] | 13.0 [8.66 to 17.28]
Statistical Analysis 1: Comparison: Sodium Oxybate 1.5 Grams (A) vs Sodium Oxybate 3 Grams (B); Test type: Superiority or Other; p = 0.013, ANOVA
Statistical Analysis 2: Comparison: Sodium Oxybate 1.5 Grams (A) vs Placebo (C); Test type: Superiority or Other; p = 0.713, ANOVA
Statistical Analysis 3: Comparison: Sodium Oxybate 3 Grams (B) vs Placebo (C); Test type: Superiority or Other; p = 0.038, ANOVA

ADVERSE EVENTS:
Arm/Group | Sodium Oxybate 1.5 Grams (A) | Sodium Oxybate 3 Grams (B) | Placebo (C)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 5/20 | 12/20 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oxybate 1.5 Grams (A) (N=20) | Sodium Oxybate 3 Grams (B) (N=20) | Placebo (C) (N=19)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (3) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling Drunk (General disorders) | 2 (2) | 5 (5) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Feeling Abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other